CLINICAL TRIAL: NCT02533388
Title: Effects of Transcutaneous Electrical Acupoint Stimulation on the Stress Response During Extubation After General Anesthesia in Elderly Patients Undergoing Elective Supratentorial Craniotomy
Brief Title: Effects of TEAS on Stress Response During Extubation of General Anesthesia in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, resident doctor, Shengjing Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TEAS on stress
Record Dates: First submitted 2015-06-04; First posted 2015-08-26 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Stress
Keywords: transcutaneous electrical acupoint stimulation; stress response
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrical acupoint stimulation (Experimental): Electrical acupoint stimulation at the Hegu (LI4), Neiguan (PC6), Lieque (LU7), Chize (LU5), Futu (LI18) and Renying (ST9) acupoints, Stimulus frequency was an alternate dense-disperse frequency of 2/10 Hz ( 2 Hz for 10 s and 10 Hz for 5 s). The optimal intensity ranged from 6-15 mA, which was adjusted to maintain a slight twitching of the regional muscles according to individual maximum tolerance.
  Interventions: Device: Hwato Electronic Acupuncture Treatment Instrument
- Sham stimulation (Sham Comparator): Sham stimulation only connected to the apparatus, but electronic stimulation was not applied.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Hwato Electronic Acupuncture Treatment Instrument — Thirty minutes prior to the induction of anaesthesia, the patients in the TEAS group started to receive TEAS by a stimulator (Hwato Electronic Acupuncture Treatment Instrument, model No.: SDZ-II, Suzhou Medical Appliances Co., Ltd., Suzhou, China) to the right hand, forearm and neck by an experienced acupuncturist at the Hegu (LI4), Neiguan (PC6), Lieque (LU7), Chize (LU5), Futu (LI18) and Renying (ST9) acupoints. TEAS was peformed with an alternate dense-disperse frequency of 2 and10 Hz ( 2 Hz for 10 s and 10 Hz for 5 s). The optimal intensity ranged from 6-15 mA, The stimulus continued until 5 min before the end of surgery.
  Arms: Electrical acupoint stimulation
Device: Placebo — The patients in the Sham group were also connected to the apparatus, but electronic stimulation was not applied.
  Arms: Sham stimulation

SUMMARY:
Elderly patients have an increased risk of stress responses during extubation after general anaesthesia for an elective supratentorial craniotomy. How to decrease the stress responses during extubation after general anaesthesia remains challenging for the anaesthesiologist. In this study, we aimed to investigate whether transcutaneous electrical acupoint stimulation (TEAS) might decrease the stress responses and improve the quality of recovery in the elderly patients who underwent elective supratentorial craniotomy under general anaesthesia.

DETAILED DESCRIPTION:
A total of 100 elderly patients scheduled for elective supratentorial craniotomy under propofol-remifentanil total intravenous anaesthesia were randomly divided to either TEAS group (received stimulation at LI4, PC6, LU7, LU5, LI18 and ST9 acupoints, 2/10Hz, 6-15 mA) or Sham group (received no stimulation). The primary outcomes were the haemodynamic parameters and plasma concentrations of epinephrine (E), norepinephrine (NE) and cortisol (Cor). The secondary outcomes were the consumption of remifentanil and propofol, the time from discontinuation of anesthetics to extubation and reorientation, extubation quality score, the quality of postoperative recovery and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* ASA Ⅱ～Ⅲ
* aged 60-70years
* scheduled for elective supratentorial craniotomy under general anaesthesia

Exclusion Criteria:

* past or current history of cardiovascular and/or cerebrovascular diseases
* diabetes
* pre-existing liver, lung or kidney dysfunction
* psychiatric disorders
* potentially difficult airway
* previous acupuncture treatment
* infection at the stimulus sites

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in Non-invasive arterial blood pressure | Before the onset of TEAS,prior to induction, at the end of surgery, immediately after extubation, and 5 and 10 min after extubation
  Non-invasive arterial blood pressure was recorded before the onset of TEAS,prior to induction, at the end of surgery, immediately after extubation, and 5 and 10 min after extubation
Change in plasma concentrations of epinephrine | Before the onset of TEAS,prior to induction, at the end of surgery, immediately after extubation, and 5 and 10 min after extubation
  plasma concentrations of epinephrine was recorded before the onset of TEAS,prior to induction, at the end of surgery, immediately after extubation, and 5 and 10 min after extubation
Change in mean arterial blood pressure | Before the onset of TEAS,prior to induction, at the end of surgery, immediately after extubation, and 5 and 10 min after extubation
  Mean arterial blood pressure was recorded before the onset of TEAS,prior to induction, at the end of surgery, immediately after extubation, and 5 and 10 min after extubation
Change in heart rate | Before the onset of TEAS,prior to induction, at the end of surgery, immediately after extubation, and 5 and 10 min after extubation
  Heart rate was recorded before the onset of TEAS,prior to induction, at the end of surgery, immediately after extubation, and 5 and 10 min after extubation
Change in norepinephrine | Before the onset of TEAS,prior to induction, at the end of surgery, immediately after extubation, and 5 and 10 min after extubation
  Norepinephrine was recorded before the onset of TEAS,prior to induction, at the end of surgery, immediately after extubation, and 5 and 10 min after extubation
Change in cortisol | Before the onset of TEAS,prior to induction, at the end of surgery, immediately after extubation, and 5 and 10 min after extubation
  Cortisol was recorded before the onset of TEAS,prior to induction, at the end of surgery, immediately after extubation, and 5 and 10 min after extubation

SECONDARY OUTCOMES:
Postoperative quality of recovery assessed by Quality of Recovery-40 questionnaire(QoR-40) | From discontinuation of anaesthetic drugs to 24 h after surgery
the time to extubation,the time to reorientation | From discontinuation of anaesthetic drugs to 24 h after surgery
the quality of extubation was evaluated by a 5-point Extubation Quality Score | From discontinuation of anaesthetic drugs to 24 h after surgery
The total amount of remifentanil that used throughout the surgery | From discontinuation of anaesthetic drugs to 24 h after surgery
The total amount of propofol that used throughout the surgery | From discontinuation of anaesthetic drugs to 24 h after surgery
Postoperative complications,like cough,agitation,nausea and vomiting | From discontinuation of anaesthetic drugs to 24 h after surgery
  Cough was assessed using a four-point scale；Agitation was evaluated using the Ricker Sedation-Agitation Scale；Nausea was defined as the patient complained of an unpleasant sensation with the urgency to vomit. Vomiting was defined as the forceful expulsion of gastric contents from the patient's mouth.

CONTACTS AND LOCATIONS:
Overall Officials: Junchao Zhu, doctor, Study Director — professor
Locations (1):
- Shengjing hospital of China medical university, Shenyang, Liaoning, China